CLINICAL TRIAL: NCT03246633
Title: Perceptual Training to Improve Early Detection of Melanoma by Future Healthcare Providers: to Accuarate Triage of Benign vs. Malignant Pigmented Skin Lesions
Brief Title: Perceptual Expertise Training for Triage of Moles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00205548
Record Dates: First submitted 2017-07-28; First posted 2017-08-11 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Lesion; Pigment; Diagnostic Self Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perceptual Training (Other): Single-Arm study, all participants will receive educational training via online modules and will be assessed after completion of the training.
  Interventions: Other: Perceptual Training

INTERVENTIONS:
Other: Perceptual Training — Participants will assess skin lesions before and after completion of an online/mobile course that has the goal of learning to triage pigmented lesions as benign or malignant. Participants will also help evaluate the usability and effectiveness of the course by completing a questionnaire after completion of the course.

SUMMARY:
The aim of this study is to assess a novel educational mobile and online application which will use images of pigmented skin lesions with question prompts to train future medical providers to more accurately detect malignant lesions.

The hypothesis of this study is that this new educational tool will result in higher melanoma detection rates among future providers.

DETAILED DESCRIPTION:
Primary Objective: To design an online and mobile course in which participants will learn to triage pigmented lesions as benign or malignant. The course will use images and question prompts to train users in pattern recognition with the goal of increased diagnostic accuracy.

Secondary Objective: To assess the effectiveness of this course. Students will be asked to rank their confidence when answering questions at the end of each module and confidence over time will be tracked. Students will also be asked to complete a post-course survey which will include an externally validated, 10 question usability scale. Responses will be standardized and compared across participants.

The study will take place at Northwestern University Feinberg School of Medicine over a 2 year time course. Initially, participants will assess the diameter of pigmented lesions with and without a ruler incorporated in the image of a pigmented lesion that contains at least one hair (Phase 1). Next, participants will be asked to complete an online/mobile course with the goal of learning to triage pigmented lesions as benign or malignant. (Phase 2) (Figure 1) These will be accessed on personal smart phones and/or computers. The course will consist of four modules of increasing difficulty. These modules will be completed in (4) 20 minute sessions over the course of 2 weeks. Each module will pair 4 images of benign lesion with 4 images of melanomas. Each sequential module will incorporate one new type of benign lesion as well as re-introduced images that were triaged incorrectly in previous modules.

At the end of each module, participants will be asked to rate their confidence in answering triaging lesions on a scale of 1-10. The change in confidence rating between Module 1 and 4 will be tracked. Students will also be asked to answer a post-test questionnaire designed to assess: i) the usability of this course ii) effectiveness of this course in helping students triage benign and malignant lesions. Usability will be assessed with the System Usability Scale. Effectiveness of the course will be assessed with questions tailored to assess the specific learning objectives.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Phase 1

Study participants must:

1. be over the age of 18
2. be currently a medical student , dermatology resident or member of the dermatology faculty at Northwestern University Feinberg School of Medicine
3. able to consent

   Inclusion Criteria for Phase 2

   Study participants must:
4. be over the age of 18
5. be currently enrolled in an MD or PA course at Northwestern University Feinberg School of Medicine
6. able to consent
7. have internet access
8. own and be able to use a smart phone
9. be willing to participate in two online surveys before and after each simulation

Exclusion Criteria:

Exclusion Criteria for Phases 1 and 2

Participants will be excluded if:

1. Not over 18 years of age
2. Do not have internet access
3. Do not have smart phone access
4. Are not currently enrolled as MD or PA students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Usability of Course | 18 months
  Usability will be assessed with the System Usability Scale, a widely accepted and validated scale to assess consumer satisfaction with new products

SECONDARY OUTCOMES:
Effectiveness of Course | 18 months
  Effectiveness of the course will be assessed with quiz requiring a benign or malignant decision about each image presents

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Society, A.C. Melanoma Skin Cancer. 2016.
- [Background] Reed KB, Brewer JD, Lohse CM, Bringe KE, Pruitt CN, Gibson LE. Increasing incidence of melanoma among young adults: an epidemiological study in Olmsted County, Minnesota. Mayo Clin Proc. 2012 Apr;87(4):328-34. doi: 10.1016/j.mayocp.2012.01.010. PMID 22469345
- [Background] Aviles-Izquierdo JA, Molina-Lopez I, Rodriguez-Lomba E, Marquez-Rodas I, Suarez-Fernandez R, Lazaro-Ochaita P. Who detects melanoma? Impact of detection patterns on characteristics and prognosis of patients with melanoma. J Am Acad Dermatol. 2016 Nov;75(5):967-974. doi: 10.1016/j.jaad.2016.07.009. Epub 2016 Sep 16. PMID 27645105
- [Background] Summaries for patients. Screening for skin cancer: U.S. Preventive Services Task Force recommendation. Ann Intern Med. 2009 Feb 3;150(3):I40. doi: 10.7326/0003-4819-150-3-200902030-00003. No abstract available. PMID 19189902
- [Background] Society, A.C. Skin Exams. 2016.
- [Background] Thomas L, Tranchand P, Berard F, Secchi T, Colin C, Moulin G. Semiological value of ABCDE criteria in the diagnosis of cutaneous pigmented tumors. Dermatology. 1998;197(1):11-7. doi: 10.1159/000017969. PMID 9693179
- [Background] Scope A, Dusza SW, Halpern AC, Rabinovitz H, Braun RP, Zalaudek I, Argenziano G, Marghoob AA. The "ugly duckling" sign: agreement between observers. Arch Dermatol. 2008 Jan;144(1):58-64. doi: 10.1001/archdermatol.2007.15. PMID 18209169
- [Background] Herschorn A. Dermoscopy for melanoma detection in family practice. Can Fam Physician. 2012 Jul;58(7):740-5, e372-8. PMID 22859635
- [Background] Brochez L, Verhaeghe E, Bleyen L, Naeyaert JM. Diagnostic ability of general practitioners and dermatologists in discriminating pigmented skin lesions. J Am Acad Dermatol. 2001 Jun;44(6):979-86. doi: 10.1067/mjd.2001.113442. PMID 11369910
- [Background] Wender RC. Barriers to effective skin cancer detection. Cancer. 1995 Jan 15;75(2 Suppl):691-8. doi: 10.1002/1097-0142(19950115)75:2+3.0.co;2-g. PMID 7804996
- [Background] Cassileth BR, Clark WH Jr, Lusk EJ, Frederick BE, Thompson CJ, Walsh WP. How well do physicians recognize melanoma and other problem lesions? J Am Acad Dermatol. 1986 Apr;14(4):555-60. doi: 10.1016/s0190-9622(86)70068-6. PMID 3958271
- [Background] Oliveria SA, Heneghan MK, Cushman LF, Ughetta EA, Halpern AC. Skin cancer screening by dermatologists, family practitioners, and internists: barriers and facilitating factors. Arch Dermatol. 2011 Jan;147(1):39-44. doi: 10.1001/archdermatol.2010.414. PMID 21242390
- [Background] Garg A, Wang J, Reddy SB, Powers J, Jacob R, Powers M, Biello K, Cayce R, Savory S, Belazarian L, Domingues E, Korzenko A, Wilson L, Grant-Kels JM, George P, Robinson-Bostom L, Trotter SC, Geller AC. The Integrated Skin Exam film: an educational intervention to promote early detection of melanoma by medical students. J Am Acad Dermatol. 2014 Jan;70(1):115-9. doi: 10.1016/j.jaad.2013.09.028. Epub 2013 Nov 9. PMID 24220723
- [Background] Lofgreen S, Lehrer M, Bennett P, Garg A, Dunnick CA. Integrating The Integrated Skin Exam film into medical education. Dermatol Online J. 2016 Nov 15;22(11):13030/qt5pk3n658. PMID 28329558
- [Background] Eide MJ, Asgari MM, Fletcher SW, Geller AC, Halpern AC, Shaikh WR, Li L, Alexander GL, Altschuler A, Dusza SW, Marghoob AA, Quigley EA, Weinstock MA; INFORMED (INternet course FOR Melanoma Early Detection) Group. Effects on skills and practice from a web-based skin cancer course for primary care providers. J Am Board Fam Med. 2013 Nov-Dec;26(6):648-57. doi: 10.3122/jabfm.2013.06.130108. PMID 24204061
- [Background] Jain N, Anderson MJ, Patel P, Blatt H, Davis L, Bierman J, McGaghie W, Brucker JB, Martini M, Robinson JK. Melanoma simulation model: promoting opportunistic screening and patient counseling. JAMA Dermatol. 2013 Jun;149(6):710-6. doi: 10.1001/jamadermatol.2013.2882. PMID 23552462
- [Background] Brooke, J., SUS: A